CLINICAL TRIAL: NCT01719822
Title: Physical Activity Augmentation Using Pedometers During Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012LF002H
Record Dates: First submitted 2012-07-20; First posted 2012-11-01 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic
Keywords: Treatment Outcome [E01.789.800]; Rehabilitation [N02.421.784]; Physical Fitness [I03.621]; Lung Diseases, Obstructive [C08.381.495]; Pulmonary Disease, Chronic Obstructive [C08.381.495.389]; Bronchitis, Chronic [C08.381.495.389.500]
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Lung Diseases; Bronchitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Standard 8-week pulmonary rehabilitation programme with 2 supervised sessions per week and a written home exercise plan/diary.
- Intervention (Experimental): Standard 8-week pulmonary rehabilitation programme with 2 supervised sessions per week. In addition they will receive a pedometer with a daily step count target set by a physiotherapist and a written home exercise plan/diary.
  Interventions: Device: Yamax Digi-Walker CW-700

INTERVENTIONS:
Device: Yamax Digi-Walker CW-700 — A pedometer with a daily step count target set by a physiotherapist.
  Arms: Intervention

SUMMARY:
Patients with chronic lung diseases such as Chronic Obstructive Pulmonary Disease (COPD), who perform regular physical activity, have improved health and wellbeing compared with those who do little exercise. The purpose of the study is to evaluate whether the use of a simple pedometer (step counter) to set targets for daily physical activity can encourage COPD patients referred for an 8-week pulmonary exercise based programme (PR) to be more active. The investigators also want to know whether the use of pedometers during PR can improve adherence, self-management and outcome in COPD.

ELIGIBILITY:
Inclusion Criteria:

* All patients with COPD

Exclusion Criteria:

* Any patient in whom mobility and lower limb function have been significantly affected by a neuromuscular disease, severe peripheral vascular disease or amputation
* Any patient whom the chief investigator feels it is unsafe to exercise (eg. unstable cardiac disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline of time spent in at least moderate physical activity (3>METS equivalent) | 8 weeks

SECONDARY OUTCOMES:
Change from baseline of Incremental Shuttle Walk | 8 weeks
Change from baseline of Chronic Respiratory Disease Questionaire (CRDQ) | 8 weeks
Change from baseline of Medical Outcomes Survey Short Form 36 item questionaire SF-36 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MRCP, PhD, Principal Investigator — Respiratory Biomedical Research Unit, Royal Brompton & Harefield NHS Foundation Trust and Imperial College London
Locations (1):
- Harefield Hospital, Middlesex, United Kingdom

REFERENCES:
- [Background] Butler L, Furber S, Phongsavan P, Mark A, Bauman A. Effects of a pedometer-based intervention on physical activity levels after cardiac rehabilitation: a randomized controlled trial. J Cardiopulm Rehabil Prev. 2009 Mar-Apr;29(2):105-14. doi: 10.1097/HCR.0b013e31819a01ff. PMID 19305235
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM. Regular physical activity modifies smoking-related lung function decline and reduces risk of chronic obstructive pulmonary disease: a population-based cohort study. Am J Respir Crit Care Med. 2007 Mar 1;175(5):458-63. doi: 10.1164/rccm.200607-896OC. Epub 2006 Dec 7. PMID 17158282
- [Derived] Nolan CM, Maddocks M, Canavan JL, Jones SE, Delogu V, Kaliaraju D, Banya W, Kon SSC, Polkey MI, Man WD. Pedometer Step Count Targets during Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2017 May 15;195(10):1344-1352. doi: 10.1164/rccm.201607-1372OC. PMID 27911566